CLINICAL TRIAL: NCT02012283
Title: Influence of Spices on Mixed Vegetable Intake Including Brassica
Brief Title: Influence of Spices on Mixed Vegetable Intake Including Brassica Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Dr. Zhaoping Li, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: VEGSPICE-12-001119
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Overcoming Resistance to Eating Cruciferous Vegetables
Keywords: spices and vegetables

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vegetable Intake with Spices Added (Experimental): Subjects consuming vegetables with mixed-spices added.
  Interventions: Other: Food consumption
- Vegetable Intake without Spices Added (Active Comparator): Subjects consuming vegetables without spice.
  Interventions: Other: Food consumption

INTERVENTIONS:
Other: Food consumption — Cooked vegetables with spices or without spices

SUMMARY:
This study is being done to determine that carefully designed spice mixtures can override any taste aversion to brassica vegetables, increase consumption of vegetable dishes which include brassica vegetables.

DETAILED DESCRIPTION:
This study is to determine the liking of vegetables, intentions to consume vegetables and differences in responses in consumption of three individual vegetables including: broccoli florets, cauliflower florets, baby spinach with and without spices added by measuring: (1) the actual intake of blanched dishes of vegetables using a modified Universal Eating Monitor when dishes are eaten plain or with added spices in random order; and (2) level of eating by baseline eating restraint using the Three Factor Eating Questionnaire (TFEQ).

This study will be conducted in healthy overweight subjects (30-60 years, Body Mass Index >25 and <30). A total of 20 subjects will be recruited (10 men and 10 women). Subjects will be further stratified by whether their level of restrained eating (10 high and 10 low restraint in each group). All participants will complete a general recruitment questionnaire which incorporates the TFEQ (Stunkard & Messick, 1985, Cappelleri 2009) along with measures of food and drink preferences and allergies. To ensure large differences in restraint between groups, subjects will be pre-selected depending on their score on the TFEQ cognitive restraint scale, with scores greater than two defined as high restraint (HR), and two or less than two as low restraint (LR). An equal number of high restraint and low restraint eaters will be tested.

Three different vegetables with or without spices given a total of 6 dishes will be tested in 6 visits per subject. The order in which each participant will be presented with the spiced or plain vegetables is randomized. Participants will be presented with a tray containing one of the three different vegetables served as a buffet in containers. As each subject ingests the dish with or without spices the rate of eating and amount eaten will be measured using a computer-based system modified from the Universal Eating Monitor.

Broccoli will be seasoned with pre-prepared spice mix containing garlic powder (0.7g), onion powder (0.7g), black pepper (0.25g) and basil leaves (0.12g); cauliflower (300g) with garlic (0.1g), dill weed (0.12g), onion (0.05g) and black pepper (0.05g); and spinach (300g) with dried chervil (0.07g), dried chives (0.13g), garlic (0.4g) and onion (0.4g).

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-60 years of age at screen.
2. BMI >25 and <30
3. In good health
4. Eat <3 serving of vegetable per day.

c. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

-

Exclusion Criteria:

1. Any history of gastrointestinal disease except for appendectomy
2. Any subject with a history of diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
3. Any subject allergic to spice or vegetables
4. Any subject who currently uses tobacco products.
5. Any subject who participates in vigorous physical activity on a regular basis.
6. Any subject who is unable or unwilling to comply with the study protocol.

   -

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li, Z. , Krak, M. , Zerlin, A. , Brahe, L. , Rheinwald-Jones, A. , Thames, G. , Zhang, Y. , Tseng, C. and Heber, D. (2015) The Impact of Spices on Vegetable Consumption: A Pilot Study. Food and Nutrition Sciences, 6, 437-444.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 11/2012 - 6/2013. The enrollment took place in a private setting the clinic located at the site.
Pre-assignment Details: Twenty subjects completed a general recruitment questionnaire were recruited. They were categorized based on their score on the Three-Factor Eating Questionnaire with score greater than 2 defined as high restraint eaters, and 2 or less defined as low restraint eaters. First Intervention was broccoli, second was cauliflower and third was spinach.
Groups:
- No Spice First, Then Spice: Subjects receiving plain vegetable, then vegetable with spices added
- Spice First, Then no Spice: Subjects receiving vegetable with mixed-spices added, then plain vegetable
Period: First Intervention
Arm/Group | No Spice First, Then Spice | Spice First, Then no Spice
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | No Spice First, Then Spice | Spice First, Then no Spice
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | No Spice First, Then Spice | Spice First, Then no Spice
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Spice First, Then Spice: Subjects consumed each vegetable without spice first and then with spice mix added
- Spice First, Then No Spice: Subjects consumed each vegetable with spice mix added first and then without spice
- Total: Total of all reporting groups
Arm/Group | No Spice First, Then Spice | Spice First, Then No Spice | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Differences Between Plain and Spiced Vegetables Intake
Description: Vegetable intake (grams) was measured while ingesting using an Universal Eating Monitor integrating a hidden weighing apparatus with specialized data collection software to analyze human eating.
Time Frame: 1 day
Population: One female low restraint eater produced irregular data that was removed from analysis population. One male high restraint eater data was removed too to obtain equal number.
Measure: Mean (Standard Deviation); unit: gram
Groups:
- Vegetable Intake With and Without Spices: The amount of vegetable consumed with or without spices.
Arm/Group | Vegetable Intake With and Without Spices
Number analyzed (Participants) | 18
gram
  Broccoli without spice | 134.1 (104.0)
  Broccoli with spice | 212.5 (155.3)
  Cauliflower without spice | 204.8 (159.2)
  Cauliflower with spice | 178.1 (119.9)
  Spinach without spice | 146.0 (167.9)
  Spinach with spice | 118.7 (105.2)
Statistical Analysis 1: Comparison: Vegetable Intake With and Without Spices; Difference between plain and spiced broccoli intake was compared; Test type: Other — paired t-test; p = 0.001, t-test, 2 sided — p<0.05 is defined as significant; Mean Difference (Final Values) = 78.4

2. Secondary Outcome: Difference in Broccoli Intake With or Without Spice Among Higher Restraint Eaters and Low Restraint Eaters
Description: Twenty subjects were categorized based on their score on the Three-Factor Eating Questionnaire with score greater than 2 defined as high restraint (HR), and 2 or less defined as low restraint (LR) eaters.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Broccoli Intake Among High Restraint Eaters: Broccoli intake with or without spices in high restraint eaters.
- Broccoli Intake Among Low Restraint Eaters: Broccoli intake with or without spices in low restraint eaters.
Arm/Group | Broccoli Intake Among High Restraint Eaters | Broccoli Intake Among Low Restraint Eaters
Number analyzed (Participants) | 9 | 9
grams
  without spice | 141.7 (122.2) | 126.4 (89.1)
  with spices added | 270.8 (186.9) | 154.2 (93.0)
Statistical Analysis 1: Comparison: Broccoli Intake Among High Restraint Eaters vs Broccoli Intake Among Low Restraint Eaters; Comparison was made to the broccoli intake with and without spices among low restraint eaters vs. the change among high restraint eaters; Test type: Other — paired t-test; p = 0.031, t-test, 2 sided — p<0.05 is defined as significant; Mean Difference (Final Values) = 101.3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over one day period for each intervention
Description: Participants were monitored and questioned regarding the occurrence and nature of any adverse experiences
Groups:
- Broccoli With Spices: Subjects consumed broccoli with spices added.
- Broccoli No Spices: Subjects consumed broccoli without spices.
- Cauliflower With Spices: Subjects consumed cauliflower with spices added.
- Cauliflower No Spices: Subjects consumed cauliflower without spices.
- Spinach With Spices: Subjects consumed spinach with spices added.
- Spinach No Spices: Subjects consumed spinach without spices.
Arm/Group | Broccoli With Spices | Broccoli No Spices | Cauliflower With Spices | Cauliflower No Spices | Spinach With Spices | Spinach No Spices
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No